CLINICAL TRIAL: NCT01056380
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of Nitazoxanide in Adults With Acute Uncomplicated Influenza
Brief Title: Study of Nitazoxanide in Adults With Acute Uncomplicated Influenza
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment during 2009-2010 flu season, new study initiated.
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM01-2027
Record Dates: First submitted 2010-01-23; First posted 2010-01-26 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Influenza
Keywords: influenza; influenza like illness
MeSH Terms: conditions — Influenza, Human | interventions — nitazoxanide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitazoxanide (Active Comparator)
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Tablet, 500 mg with food twice daily for 5 days
  Other Names: Alinia, NTZ
  Arms: Nitazoxanide
Drug: Placebo — Tablet, twice daily with food for 5 days
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This is a randomized clinical trial designed to evaluate oral nitazoxanide compared to a placebo in the treatment of acute uncomplicated influenza in adults. We hypothesize that treatment with nitazoxanide will reduce the duration of symptoms in patients with confirmed influenza infection. Secondarily, we hypothesize that treatment with nitazoxanide will reduce the complications of influenza, severity of symptoms, time lost from work, time to return to normal daily activities, and viral shedding.

DETAILED DESCRIPTION:
The study is conducted at approximately 25 sites in the United States. Subjects selected based on symptoms will be randomized to receive oral nitazoxanide or placebo twice daily for 5 days. Subjects will be monitored by daily by telephone or home visit to monitor symptoms and complications of influenza for safety and will be referred for medical care as required. Subjects will complete a diary twice daily to record the presence and severity of symptoms, ability to perform normal daily activities and time lost from work. Complications of influenza (including sinusitis, otitis, bronchitis, pneumonia, central nervous system disease) and other adverse events will be reported. Nasopharyngeal swabs will be collected at Baseline (Day 0) and Day 7 for all patients and on Days 1 through 4 for a subset of patients to test for influenza A (including novel H1N1), influenza B and 17 other respiratory viruses by RT-PCR and culture and to evaluate quantitative viral shedding. The primary analysis will be for patients with confirmed influenza, and secondary analyses will be conducted for subjects with any respiratory virus and for all treated subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Fever, respiratory symptoms and constitutional symptoms compatible with influenza infection
* Influenza A or B infection in the local community
* Onset of illness no more than 48 hours before presentation
* Willing and able to provide comply with protocol requirements

Exclusion Criteria:

* Severity of illness requiring or anticipated to require in-hospital care
* High risk of complications from influenza per IDSA (Infectious Diseases Society of America) guidelines or current CDC (Centers for Disease Control) criteria
* Females pregnant, breast-feeding or sexually active without birth control
* Vaccination for seasonal influenza or H1N1 on or after August 1, 2009
* Treatment with antiviral medication for influenza within 1 month prior to screening
* Treatment with nitazoxanide or any investigational drug within 1 month prior to screening
* Known sensitivity to nitazoxanide or any excipients
* Unable to take oral medications
* Chronic kidney or liver disease or known impaired hepatic and/or renal function
* Other pre-existing chronic infection undergoing or requiring medical therapy
* Pre-existing illness placing subject at unreasonably increased risk by participation in study
* Unlikely to comply with the requirements of this protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Rossignol, MD, PhD, Study Chair — The Romark Institute for Medical Research
Locations (1):
- Health Sciences Research Center at Asthma and Allergy Associates, P.C., Elmira, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 11 primary care health centers throughout the United States in the last months of the 2009/2010 flu season
Groups:
- Nitazoxanide: Nitazoxanide : Tablet, 500 mg with food twice daily for 5 days
- Placebo: Placebo : Tablet, twice daily with food for 5 days
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 37 | 42
Completed | 35 | 39
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 37 | 42 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 42 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (14.4) | 37.9 (13.3) | 38.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 37 | 42 | 79

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of All Clinical Symptoms of Influenza (Subjects With Confirmed Influenza Infection)
Time Frame: Up to 28 days
Population: All subjects with laboratory confirmed influenza who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 3 | 3
hours | 55.0 [12 to 176] | 91.5 [70 to 178]

2. Secondary Outcome: Time to Resolution of All Clinical Symptoms of Influenza (Subjects Infected With Any Respiratory Virus)
Time Frame: Up to 28 days
Population: All subjects with any laboratory confirmed viral infection who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 20 | 22
hours | 118.0 [80 to 157] | 88.8 [70 to 139]

3. Secondary Outcome: Time to Resolution of All Clinical Symptoms of Influenza (All Treated Subjects)
Time Frame: Up to 28 days
Population: All subjects who received at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 37 | 40
hours | 119.8 [72 to 169] | 102.6 [69 to 141]

4. Secondary Outcome: Time to Return to Normal Daily Activity (Subjects With Confirmed Influenza)
Time Frame: Up to 28 days
Population: All subjects with laboratory confirmed influenza who received at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 3 | 3
hours | 48.5 [31 to 176] | 57.5 [21 to 128]

5. Secondary Outcome: Overall Severity of Disease Score
Description: Subjects recorded a severity score for 10 flu symptoms on a 0-3 scale BID for 7-14 days.The severity score for each symptom was multiplied by the number of hours scored at that severity for the entire time the subject maintained a diary (a sneezing score of 1 for 12 hours and 0 for 10 hours =1*12 + 0*10=12). This is symptom severity score*hours.Symptom severity score*hours for each of the symptoms were added for an overall symptom severity score*hours (if symptom severity score*hours for 10 symptoms were 12, 10, 9, 8, 7, 10, 10, 10, 5, 5, overall symptom severity score*hours=86).Overall symptom severity score*hours were divided by the number of hours that the subject kept a diary for a standardized continuous measure of severity of the course of illness (if overall symptom severity score*hours=86 and the subject maintained a diary for 100 hours Overall Severity of Disease Score=0.86). Overall Severity of Disease Score can range 0-30 with higher scores indicating more severe symptoms.
Time Frame: Up to 14 days
Population: All subjects with laboratory confirmed influenza who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: overall severity score
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 3 | 3
overall severity score | 5.4 (3.3) | 6.2 (3.6)

6. Secondary Outcome: Time Lost From Work (Subjects With Confirmed Influenza)
Time Frame: Up to 28 days
Population: All subjects with laboratory confirmed influenza who received at least one dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 3 | 3
hours | 3.64 [-0.04 to 7.32] | 4.36 [-0.70 to 9.42]

7. Secondary Outcome: Complications of Influenza Including Secondary Illnesses, Antibiotic Use and Hospitalizations (Subjects With Confirmed Influenza)
Time Frame: Up to 28 days
Population: All subjects with laboratory confirmed influenza who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

8. Secondary Outcome: Time to Cessation of Viral Shedding (Subjects With Confirmed Influenza)
Time Frame: 28 days
Population: All subjects with laboratory confirmed influenza enrolled in the intensive virologic follow up substudy who received at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 1 | 2
hours | 95.5 [95.5 to 95.5] | 83.3 [72 to 95]

9. Secondary Outcome: Change in Influenza Virus Titer Assessed by Quantitative RT-PCR (Subjects With Confirmed Influenza)
Time Frame: 4 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Quantitative PCR RNA Copies
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 1 | 2
Quantitative PCR RNA Copies
  Baseline | 0 (0) | 0 (0)
  Day 2 | 0 (0) | -175183057 (373069697)
  Day 3 | 0 (0) | -176973304 (374681622)
  Day 4 | 0 (0) | -176946354 (375523235)

ADVERSE EVENTS:
Arm/Group | Nitazoxanide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/42
Other Adverse Events (participants affected / at risk) | 9/37 | 6/42
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=37) | Placebo (N=42)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (3) | 4 (5) — Abdominal distension, Abdominal pain upper, Diarrhea, Dysgeusia, Nausea, Oropharyngeal pain
General disorders and administration site conditions (General disorders) | 1 (1) | 1 (1) — Malaise, Pyrexia
Infections and infestations (Ear and labyrinth disorders) | 2 (2) | 2 (3) — Ear infection, Sinusitis
Muscoloskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Arthralgia
Nervous system disorders (Nervous system disorders) | 1 (1) | 2 (2) — Headache
Renal and urinary disorders (Renal and urinary disorders) | 3 (3) | 0 (0) — Chromaturia, Pollakiuria
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Epididymitis
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) — Cough, Dyspnoea, Productive cough

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Presentation and/or publication is encouraged provided the Sponsor is notified in advance and given the opportunity to review the manuscript or abstract 30 days prior to its submission for presentation at a scientific meeting or for publication in a scientific journal. The investigators will have complete autonomy regarding the content and wording including the decision of whether or not to publish.